CLINICAL TRIAL: NCT05396430
Title: Early Recovery After Cesarean Delivery: Duration of Urinary Catheter Treatment
Brief Title: Duration of Urinary Catheter Treatment After Cesarean Delivery Under Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Women's Hospital HUS (Other)
Responsible Party: Principal Investigator, Antti Vaananen, Principal investigator, Women's Hospital HUS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tutkimussuunnitelma25032022
Record Dates: First submitted 2022-05-27; First posted 2022-05-31 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Urinary Retention; Cesarean Section Complications
MeSH Terms: conditions — Urinary Retention | interventions — Urinary Catheters

STUDY DESIGN:
Intervention Model Description: The parturients are randomized into 3 different treatment arms with different duration of planned urinary catheter treatment
Masking Description: Masking is not applicable, duration of urinary catheter treatment is decided at the time of surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Urinary catheter 8 hours (Experimental): The urinary cathter is to be removed at 8 hours after the end of surgery
  Interventions: Device: Urinary catheter
- Urinary catheter 10 hours (Experimental): The urinary cathter is to be removed at 10 hours after the end of surgery
  Interventions: Device: Urinary catheter
- Urinary catheter 12 hours (Active Comparator): The urinary cathter is to be removed at 12 hours after the end of surgery
  Interventions: Device: Urinary catheter

INTERVENTIONS:
Device: Urinary catheter — Duration of planned urinary cathterization following cesarean delivery

SUMMARY:
In this study a total of 150 parturients undergoing cesarean delivery under spinal anesthesia will be randomized to have their urinary catheters kept in place for 8, 10 or 12 hours. The incidence of urinary retention and interventions needed for any potential urinary retention will be assessed.

DETAILED DESCRIPTION:
In this study a total of 150 parturients undergoing cesarean delivery under spinal anesthesia will be randomized to have their urinary catheters kept in place for 8, 10 or 12 hours. The incidence of urinary retention and interventions needed for any potential urinary retention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* After informed consent, signed the participation form (volunteered for the study)
* Cesarean section
* Spinal anesthesia

Exclusion Criteria:

* Prior neuraxial analgesia (epidural or spinal) for attempted labour

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Success of spontaneous voiding of bladder | 6-12 hours after removal of the urinary catheter
  Assessed by ultrasound bladder scanner after attempted voiding of the bladder

SECONDARY OUTCOMES:
Amount of residual urine in the bladder | 6-12 hours after removal of the urinary catheter
  Assessed by ultrasound
Need for standard in-house medications to help spontaneous voiding of the bladder | 6-12 hours after removal of the urinary catheter
  Amount of medicines given
Need for re-cathterization of the bladder | 6-12 hours after removal of the urinary catheter

CONTACTS AND LOCATIONS:
Locations (1):
- HUS/Women's hospital dept of obstetrics, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No